CLINICAL TRIAL: NCT03498547
Title: Comparison of Caudal Block and Saddle Block on Anorectal Surgery
Brief Title: Caudal Block,Saddle Block, Anorectal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, tahsin şimşek, specialist doctor, Kocaeli Derince Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-384
Record Dates: First submitted 2018-04-06; First posted 2018-04-13 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Anorectal Disorder
Keywords: caudal block; saddle block
MeSH Terms: conditions — Rectal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal Block (Active Comparator): For the caudal block, sacral horns are palpated and sacral hiatus and epidural area will be determined at S4-S5 level through ultrasonography. The 20 G adult caudal needle will then be placed to the caudal epidural space and 25 mL bupivacaine at a concentration of 0.5% will be applied in the prone Jack-Knife position with resistance loss.
  Interventions: Procedure: caudal block
- Saddle Block (Active Comparator): In the saddle block group hyperbaric bupivacaine at a dose of 7 mg will be given to the intrathecal space after a 25 G quincke spinal needle is inserted with ultrasonography guidance between L4-L5 vertebral disc and clear cerebrospinal fluid is seen. The patient will be placed in sitting position for 5 minutes.
  Interventions: Procedure: saddle block

INTERVENTIONS:
Procedure: caudal block — For the caudal block, sacral horns are palpated and sacral hiatus and epidural area will be determined at S4-S5 level through ulştrasonography. The 20 G adult caudal needle will then be placed to the caudal epidural space and 25 mL bupivacaine at a concentration of 0.5% will be applied in the prone Jack-Knife position with resistance loss.
  Arms: Caudal Block
Procedure: saddle block — In the saddle block group hyperbaric bupivacaine at a dose of 7 mg will be given to the intrathecal space after a 25 G quincke spinal needle is inserted with ultrasonographyguidance between L4-L5 vertebral disc and clear cerebrospinal fluid is seen. The patient will be placed in sitting position for 5 minutes.
  Arms: Saddle Block

SUMMARY:
Anorectal surgery includes pilonidal sinus, hemorrhoidectomy, anal fissure, and anal fistula operations. Various surgical and anesthetic techniques have been used to increase the level of analgesia in perioperative period and decrease the length of stay in the hospital. In this study, investigators investigate the effects of routinely applied anesthesia techniques during anorectal surgery, caudal block and saddle block, on patients' perioperative hemodynamic values, sensory and motor block levels, and postoperative pain scores.

DETAILED DESCRIPTION:
Anorectal surgery includes pilonidal sinus, hemorrhoidectomy, anal fissure, and anal fistula operations. Various surgical and anesthetic techniques have been used to increase the level of patients perioperative analgesia and decrease the length of stay in the hospital.

Spinal Saddle block anesthesia applications are performed while the patient is in the sitting position. Local anesthetic is given into the intrathecal space and it is aimed to localize the applied agent around the hip and anorectal region with the effect of gravity. Thus, sufficient level of anesthesia required during perianal region surgery and stable patient hemodynamics is provided. Caudal block is widely used in both adults and pediatric patients for intraoperative anesthesia and chronic pain management. Sacral hyperattenuation is performed to reach the epidural space, a local anesthetic agent is given to the epidural space, it is accepted as an easy and safe method and therefore it is frequently used in anorectal surgeons.

In this study, investigators investigate the effects of routinely applied anesthesia techniques during anorectal surgery, caudal block and saddle block, on patients' perioperative hemodynamic values, sensory and motor block levels, and postoperative pain scores. Elective anorectal surgery planned 100 patients between the 18-60 ages. The risk of anesthesia in patients will be determined by ASA (American Society Of anesthesiologists), ASA1 or ASA 2 risk group will be included after informed consents are approved.

Patient electrocardiogram (ECG), peripheral oxygen saturation (SpO2), non-invasive blood pressure monitor will be performed in the operation room. Baseline hemodynamic-vital parameters of the patients will be recorded. Patients undergoing caudal and saddle blocks, will be compared as two randomized groups.

In the saddle block group hyperbaric bupivacaine at a dose of 7 mg will be given to the intrathecal space after a 25 G quincke spinal needle is inserted with ultrasonography guidance between L4-L5 vertebral disc and clear cerebrospinal fluid is seen. The patient will be placed in sitting position for 5 minutes.

For the caudal block, sacral horns are palpated and sacral hiatus and epidural area will be determined at S4-S5 level through ultrasonography. The 20 G adult caudal needle will then be placed to the caudal epidural space and 25 mL bupivacaine at a concentration of 0.5% will be applied in the prone Jack-Knife position with resistance loss. Sensory and motor block level, heart rate (HR), systolic arterial pressure (SAB), diastolic arterial pressure (DAB), mean arterial pressure (OAB) and SpO2 levels will be measured every 5 minutes until the end of the operation. Sensory block level will be evaluated with "pinprick" test. Motor block level will be evaluated by using Modified Bromage Scale (0 = no paralysis, thigh, leg and foot can be removed, 1 = unable to move the thigh, move the knee,2 = cannot move the knee, can move the ankle, 3 = cannot move the lower extremities at all) Once sensory block level is reached to the L3 level the surgical procedure will begin.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old patients
* ASA 1-2 patients
* Patients who will undergo anorectal surgery

Exclusion Criteria:

* Having known hypersensitivity to amide type local anesthetics
* Patients with contraindications to central block (caudal, saddleblock): use of anticoagulant medication, local infection in the intervention site, increased intracranial pressure, severe aortic and / or mitral valve stenosis, ischemic hypertrophic subaortic stenosis,
* Patients who do not accept regional anesthesia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
The goal is to create adequate anesthesia for the surgeon to be painless | Sufficient anesthesia is expected within 30 minutes after the anesthetic agent is applied
  When anesthetic agent is administered, the formation of sensory block at level lumbar 3 vertabra will be considered as an adequate level of anesthesia

SECONDARY OUTCOMES:
The goal is to provide pain relief in the postoperative period | Postoperative follow-up for analgesia is 24 hours.
  Pain measurement will be done with a visual analogue scale for 24 hours from the end of the operation. Visual Analog Scale (VAS) is used to convert some numerically unmeasured values into numeric values. Two extremes of a 100 mm line are to be assessed on two extremes and the patient is asked to indicate on the line where his situation is appropriate by drawing a line or placing a point or pointing. For example, for pain; no pain on one tip = 0, very severe pain = 100 on the other tip, and the patient marks his / her current state on this line. According to this chart, values of 50 mm and above are adversely affecting patient comfort. Patients with visual analog scale values above 50 mm will be intervened by making analgesic drugs.

CONTACTS AND LOCATIONS:
Overall Officials: tahsin şimşek, MD, Principal Investigator — KOCAELİ DERİNCE EĞİTİM VE ARAŞTIRMA HASTANESİ; kemal tolga saracoğlu, MD, Study Director — KOCAELİ DERİNCE EĞİTİM VE ARAŞTIRMA HASTANESİ
Locations (2):
- Turkey (Türkiye) (2):
  - Derince Eğitim Ve Araştırma Hastanesi, Kocaeli, Derince
  - Şimşek, Kocaeli, Derince